CLINICAL TRIAL: NCT06715293
Title: A Prospective Study to Evaluate the Diagnostic Performance of a Wireless Optical Sensor Capsule in Detection of Upper Gastrointestinal Bleeding
Brief Title: A Study to Evaluate the Performance of a Wireless Optical Sensor Capsule in Detection of UGIB
Acronym: Hemopill-Pro
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2024.181
Record Dates: First submitted 2024-11-22; First posted 2024-12-04 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Melena; Gastrointestinal Bleeding; Hematemesis
Keywords: GIB; gastrointestinal bleeding; melena; per rectal bleeding; coffee ground vomiting; hematemesis
MeSH Terms: conditions — Melena; Gastrointestinal Hemorrhage; Hematemesis

STUDY DESIGN:
Intervention Model Description: All patient will swallow Hemopill to observe the presence of active bleeding or potential bleeding source
Who Masked: Outcomes Assessor
Masking Description: Endoscopists will be blinded from the Hemopill capsule examination results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemopill to detect the presence of active bleeding in the upper GI tract (Experimental): Hemopill to detect the presence of active bleeding in the upper GI tract
  Interventions: Device: Hemopill; Procedure: OGD
- OGD to diagnose and treat active beleeding in the upper GI tract (Active Comparator): ogd will be performed to compare the results with that of the hemopill
  Interventions: Device: Hemopill; Procedure: OGD

INTERVENTIONS:
Device: Hemopill — Hemopill will be swallowed to detect the presence of active bleeding in the upper GI tract
Procedure: OGD — OGD will be performed to compare the results of the hemopill

SUMMARY:
Upper gastrointestinal bleeding (UGIB) is a common and potentially lethal medical emergency, which requires hospitalization and healthcare resources. Despite the changing epidemiology and advancement of endoscopic therapy in the recent decade, the all-cause mortality of UGIB remains high (>2%). An accurate risk stratification is necessary to triage patients into low- or high-risk groups, in order to inform clinicians for the necessity and timing of urgent endoscopy. However, existing pre-endoscopy risk scores, such as the Glasgow-Blatchford score (GBS), Rockall score and AIMS65 score, are suboptimal in predicting relevant clinical outcomes. An alternative strategy for risk stratification is urgently warranted in patients with UGIB to guide the next step of management.

In a pre-clinical study, the sensitivity and specificity of HemoPill® prototype were 95% and 87.5% respectively, when the sensors were positioned close to the bleeding point. Furthermore, several human clinical studies have proven the feasibility and accuracy of HemoPill® in healthy volunteers and patients with suspected UGIB. Capsule ingestion was well tolerated with no device-related adverse event or capsule retention. All patients with negative HI were found to have no active endoscopic bleeding (true negative, 100%, 17/17). In patients with bleeding >20ml, true positive HI signals were detected (100%, 2/2) In a retrospective multi-center study, 61 patients with suspected UGIB were recruited to use HemoPill®. Among the capsule-positive cases, subsequent endoscopy confirmed active bleeding in 57% (20/35) of them. None of the capsule-negative patients rebled (0%, 0/25), which prevented unnecessary emergent endoscopy in 72% of them (18/25).

DETAILED DESCRIPTION:
From December 2023 to February 2024, the investigator conducted a pilot study and screened 51 adult subjects with symptoms and signs of suspected UGIB in Prince of Wales Hospital. Among them, the investigator recruited 20 eligible subjects to receive HemoPill® examination before oesophago-gastro-duodenoscopy (OGD). The overall sensitivity was 80% with a negative predictive value of 87.5%. The area-under-receiver-operating-characteristic curve was 0.633.

The pilot data demonstrated a huge potential for this novel, non-invasive, easy-to-use device as UGIB screening in the real-world. A large-scale, prospective validation study will be conducted to evaluate the diagnostic performance of the new generation HemoPill® acute capsule in UGIB.

ELIGIBILITY:
Inclusion Criteria:

1. Participants have symptoms and signs of suspected UGIB (melena, per rectal bleeding, coffee ground vomiting, prior hematemesis);
2. Participants will undergo urgent or elective OGD within 24 hours from recruitment;
3. Written consent obtained.

Exclusion Criteria:

1. Contraindications for OGD (e.g. respiratory failure, suspected perforation);
2. Contraindications for capsule endoscopy (e.g. known gastrointestinal obstruction or stricture, severe dysphagia, impaired consciousness);
3. Cardiac pacemaker or implanted electromedical devices;
4. History of gastrectomy or bowel resection;
5. Ongoing fresh hematemesis requiring emergent endoscopy;
6. Unstable hemodynamics despite adequate resuscitation requiring emergent endoscopy (i.e. systolic blood pressure <100mmHg or pulse rate >100 per minute);
7. Advanced comorbidities (defined as American Society of Anesthesiologists grade 4 or above);
8. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Presence of active bleeding | during OGD examination
  Presence of active bleeding, old blood or potential bleeding sources during OGD examination, which warrants endoscopic haemostatic treatment.

SECONDARY OUTCOMES:
Technical success rate | during OGD examination
  Technical success rate
Adverse event rate | 30days post study procedure
  Adverse event rate
Capsule retention rate | 30days post study procedure
  Capsule retention rate
Time from Hemopill acute capsule ingestion to a positive HI signal | during OGD examination
  Time from Hemopill acute capsule ingestion to a positive HI signal

CONTACTS AND LOCATIONS:
Overall Officials: Louis HS Lau, FRCP, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No